CLINICAL TRIAL: NCT01452360
Title: A Research Proposal to Set up an Integrated National Data Bank and Monitoring System and to Establish the Indicators and Risk Factors for Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yung-Ho Hsu, doctor, Taipei Medical University WanFang Hospital
Other Study IDs: 100009
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Collection of CKD patient group
- Collection of CKD high-risk group
- Collection of healthy control group

SUMMARY:
This project expects the integrated database of terminally renal ill patients combines clinical and files of Health Insurance and renal medical society database. It will provide valuable actual evidence data to quality monitoring of dialysis treatment and related academic research. Besides, using the cohort study of chronic renal disease --「epidemiologic research of chronic renal disease」, we can trace the patient continually and analysis different risk factors of chronic renal disease in Taiwan. Taken together, the results of this project --1.1「Integrate the current database of renal disease and establishment of national monitor system」and 1.2「Epidemiologic study in chronic renal disease」-- will provide the basic rules of prevention and treatment, basic research and clinic application in chronic renal disease.

DETAILED DESCRIPTION:
The main source of patient in this study sub-plan 1.2 will collect the patient from medical center in Taiwan. We assume collect 7 groups in study period -- First：【CKD stage I】. Second：【CKD stage II】. Third：【CKD stage III】. Forth：【CKD stage IV】. Fifth：【CKD stage V】. Sixth：【CKD high-risk group】. Seventh：【health control group】to study case report；Total collect 11500 people. At the same time, we collect the sample of blood and urine and personal health survey to provide the basic data base for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Collection of CKD patient group： The patients who will select into this plan are chosen from the hospital (This hospital is defined as the renal disease improving institute) in Taiwan. New case in this hospital will be collected into the CKD patient group. In order to separate those patients into five stages of CKD, we are going to calculate the glomerular filtration rate (GFR) by using the formula of GFR. Stage I -- Renal function is normally and protein was detectable slightly in urine (GFR：≧90ml/min/1.73M2). Stage II -- Slight renal function failure was observed (GFR：60~89ml/min/1.73M2). Stage III -- Moderate renal function failure (GFR：30~59ml/min/1.73M2). Stage IV -- Severe renal function failure (GFR：15~29ml/min/1.73M2). Stage V -- End stage renal disease (GFR：<15ml/min/1.73M2). The age is from fourteen to eighty-five and whatever they are male or female will be taken into this project.
2. Collection of CKD high-risk group： The CKD patient's relative will be considerately incorporated into the CKD high-risk group. If CKD patient being confirmed, their relative who had chronic disease including DM, hypertension and CVD will be chosen into CKD high-risk group. The age is from fourteen to eighty-five and whatever they are male or female. This plan will select five thousand people into CKD high-risk group.
3. Collection of healthy control group： According to the characteristic of CKD patient group, we will select the health control group carefully (paired selection of CKD patient group, 1:1). The rules of paired selection : 1. Sex 2.Age ± 5 years 3.Location -- CKD patient and health people are get from the same hospital. Health people who had no any chronic disease and required a physical checkup which get from the hospital (This hospital should be qualified to the renal disease improving institute) will be chosen into this project. Fifteen hundred people will be taken in this plan.

Exclusion Criteria:

* This plan divide into three groups：1. CKD patient group -- CKD patient group have no exclusion criteria. 2. CKD high-risk group -- CKD high-risk group exclude the patient who had renal disease. 3. Heath control group -- Heath control group exclude the patient who had any chronic disease. Test of liver residual function will exclude the patient who had allergic reactions to galactose. It will exclude the person including galactosemia patient, DM patient, pregnant woman, children and disabled people.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic kidney disease patients
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2011-05; Study Completion 2014-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Ho Hsu, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University - Shuang-Ho Hospital, Taipei, Taiwan